CLINICAL TRIAL: NCT05566808
Title: Prospective Trial Evaluation the Long-term Outcomes Associated With the Use of MTF Allograft Cartilage in Cosmetic and Reconstructive Rhinoplasty Procedures
Brief Title: Use of Allograft Cartilage in Cosmetic and Reconstructive Rhinoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTF Profile Study
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Rhinoplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Costal Cartilage Graft (Other): Patients undergoing rhinoplasty will receive autologous rib graft.
  Interventions: Other: Autologous Costal Cartilage Graft
- Costal Cartilage Allograft (Other): Patients undergoing rhinoplasty will receive costal cartilage allograft.
  Interventions: Other: Costal Cartilage Allograft.

INTERVENTIONS:
Other: Autologous Costal Cartilage Graft — Subjects undergoing either reconstructive or cosmetic rhinoplasty will choose which graft will be used in their intervention.
  Arms: Autologous Costal Cartilage Graft
Other: Costal Cartilage Allograft. — Subjects undergoing either reconstructive or cosmetic rhinoplasty will choose which graft will be used in their intervention.
  Arms: Costal Cartilage Allograft

SUMMARY:
This is a single-center, blinded, controlled trial, conducted in healthy adult subjects undergoing a reconstructive or cosmetic rhinoplasty involving the use of cartilaginous graft (either non-irradiated cartilage sheet allograft compared to autologous harvest and grafting of costal cartilage).

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo a reconstructive or cosmetic surgical procedure to alter the appearance of the nose that is anticipated to require a cartilage graft.
* Subject is willing to sign an informed consent.
* Subject is a non-smoker or has stopped smoking at least 6-weeks prior to inclusion in the study.
* Subjects must agree to forgo any treatment, medical or non-medical, to the area treated in this study, for the duration of the 1-year post-treatment evaluation period, unless there is prior approval from the investigator.

Exclusion Criteria:

* Presence of significant endocrine, immunologic, dermatologic or psychiatric abnormalities that would render the subject an inappropriate candidate for the study.
* Presence of any malignancy not considered cured in the midface area specifically (no evidence of cancer recurrence in the previous five years).
* History of radiation to the area(s) to be treated in the study.
* Subjects taking chronic steroids (injected or oral) or other immune modulators.
* Subjects with a history of skin sensitivity (dermatitis) to either the suture materials or dressings to be utilized during the course of this study.
* Subjects with skin conditions that could result in poor healing or widened scars.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Patient Outcome Assessment | Preoperative
  Subjective assessment using the Face-Q checklists and scoring for preoperative assessment.
Patient Outcome Assessment | 3 months post-operative
  Subjective assessment using the Face-Q checklists and scoring for post-operative assessments.
Patient Outcome Assessment | 6 months post-operative
  Subjective assessment using the Face-Q checklists and scoring for post-operative assessments.
Patient Outcome Assessment | 12 months
  Subjective assessment using the Face-Q checklists and scoring for post-operative assessments.

SECONDARY OUTCOMES:
Cost analysis of utilizing the different grafts as far as graft cost, operative time, re-operation, etc. | 12 months
Comparison of the overall complication rate between the MTF cartilage graft and autologous cartilage graft used during the procedures. | 12 months

OTHER OUTCOMES:
Safety: occurrence of adverse events (AEs) | 12 months
  Evaluation of the occurrence of adverse events (AEs) as documented by the treating physician during the course of treatment and follow-up visits and as reported by the subjects at each Assessment Visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States